CLINICAL TRIAL: NCT04201639
Title: Evaluating the Performance of Precision1 Daily Disposable Contact Lens in a Group of Heavy Digital Device Users
Acronym: PUG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 41694
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Refit (Experimental): Refit and dispense patient with Verofilcon A contact lenses and evaluate lens performance.
  Interventions: Device: Verofilcon A contact lenses

INTERVENTIONS:
Device: Verofilcon A contact lenses — Daily disposable silicone hydrogel contact lenses indicated for the optical correction of refractive ametropia (myopia and hyperopia)
  Other Names: Precision1™

SUMMARY:
The purpose of this study is to evaluate the performance of Precision1 DD CLs with regard to subjective symptoms (dryness, comfort, vision), lens fit and time to haze in CL wearers who identify themselves as heavy digital devices users (at least 6 hours of digital device use per day).

ELIGIBILITY:
Inclusion Criteria:

1. Is between 18 and 40 years of age (inclusive) and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Is a heavy digital device user (at least 6 hours on a typical day using any combination of digital devices such as PC, laptop, smartphone, or tablet);
5. Is a habitual wearer of daily, spherical, soft contact lenses (no bifocal or multifocal contact lenses, no extended wear or monovision, not a current wearer of Precision1 lenses) for at least 5 days/week and at least 10 hours/day during the month prior to enrollment;
6. Has a vertex corrected spherical equivalent distance refraction that ranges between -0.50D to -6.00D in each eye;
7. Has a vertex corrected refractive cylinder of no more than -1.00D cylindrical correction in each eye after vertexing to the corneal plane;
8. Demonstrates an acceptable fit and achieves best corrected visual acuity of at least 0.20 log MAR in each eye with Precision1 contact lenses;
9. Is willing to wear Precision1 CLs at least 5 days per week and 10 hours per day throughout the study;

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has any known active* ocular disease and/or infection;
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
5. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
6. Is pregnant, lactating or planning a pregnancy at the time of enrolment;
7. Is aphakic;
8. Has undergone refractive error surgery;

   * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FCOptom, Principal Investigator — Centre for Ocular Research & Education
Locations (1):
- Centre for Ocular Research & Education, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Refit
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Refit
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 32

OUTCOME MEASURES:

1. Primary Outcome: Subjective Comfort After Contact Lens Insertion
Description: Participants rate their comfort after insertion on a scale from 0 (worst) to 100 (best).
Time Frame: Dispense Visit (Day 0)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 95 [40 to 100]

2. Primary Outcome: Subjective Dryness After Contact Lens Insertion
Description: Participants rate their dryness after insertion on a scale from 0 (worst) to 100 (best).
Time Frame: Dispense Visit (Day 0)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 100 [70 to 100]

3. Primary Outcome: Subjective Rating of Clarity of Vision After Contact Lens Insertion
Description: Participants rate their clarity of vision after insertion on a scale from 0 (worst) to 100 (best).
Time Frame: Dispense Visit (Day 0)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 98 [70 to 100]

4. Primary Outcome: Subjective Comfort After Contact Lens Insertion
Description: Participants rate their comfort after insertion on a scale from 0 (worst) to 100 (best).
Time Frame: Day 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 96 [75 to 100]

5. Primary Outcome: Subjective Dryness After Contact Lens Insertion
Description: Participants rate their dryness after insertion on a scale from 0 (worst) to 100 (best).
Time Frame: Day 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 100 [80 to 100]

6. Primary Outcome: Subjective Rating of Clarity of Vision After Contact Lens Insertion
Description: Participants rate their clarity of vision after insertion on a scale from 0 (worst) to 100 (best).
Time Frame: Day 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 99 [78 to 100]

7. Primary Outcome: Subjective Comfort After Contact Lens Insertion
Description: Participants rate their comfort after insertion on a scale from 0 (worst) to 100 (best).
Time Frame: Day 7
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 98 [75 to 100]

8. Primary Outcome: Subjective Dryness After Contact Lens Insertion
Description: Participants rate their dryness after insertion on a scale from 0 (worst) to 100 (best).
Time Frame: Day 7
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 100 [80 to 100]

9. Primary Outcome: Subjective Rating of Clarity of Vision After Contact Lens Insertion
Description: Participants rate their clarity of vision after insertion on a scale from 0 (worst) to 100 (best).
Time Frame: Day 7
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 100 [80 to 100]

10. Primary Outcome: Subjective Comfort After Contact Lens Insertion
Description: Participants rate their comfort after insertion on a scale from 0 (worst) to 100 (best).
Time Frame: Day 10
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 95 [65 to 100]

11. Primary Outcome: Subjective Dryness After Contact Lens Insertion
Description: Participants rate their dryness after insertion on a scale from 0 (worst) to 100 (best).
Time Frame: Day 10
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 90 [60 to 100]

12. Primary Outcome: Subjective Rating of Clarity of Vision After Contact Lens Insertion
Description: Participants rate their clarity of vision after insertion on a scale from 0 (worst) to 100 (best).
Time Frame: Day 10
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 95 [75 to 100]

13. Primary Outcome: Subjective Comfort After Contact Lens Insertion
Description: Participants rate their comfort after insertion on a scale from 0 (worst) to 100 (best).
Time Frame: Followup visit (occurring at a single visit any day from Day 12-16)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 90 [60 to 100]

14. Primary Outcome: Subjective Dryness After Contact Lens Insertion
Description: Participants rate their comfort after insertion on a scale from 0 (worst) to 100 (best).
Time Frame: Followup visit (occurring at a single visit any day from Day 12-16)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 90 [40 to 100]

15. Primary Outcome: Subjective Rating of Clarity of Vision After Contact Lens Insertion
Description: Participants rate their comfort after insertion on a scale from 0 (worst) to 100 (best).
Time Frame: Followup visit (occurring at a single visit any day from Day 12-16)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 91 [70 to 100]

16. Primary Outcome: Subjective Comfort With Contact Lens Wear After 6 Hours of Digital Device Use
Description: Participants rate their comfort after 6 hours of digital device use on a scale from 0 (worst) to 100 (best).
Time Frame: Day 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 99 [85 to 100]

17. Primary Outcome: Subjective Dryness With Contact Lens Wear After 6 Hours of Digital Device Use
Description: Participants rate their dryness after 6 hours of digital device use on a scale from 0 (worst) to 100 (best).
Time Frame: Day 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 100 [70 to 100]

18. Primary Outcome: Subjective Rating of Vision Clarity With Contact Lens Wear After 6 Hours of Digital Device Use
Description: Participants rate their vision clarity after 6 hours of digital device use on a scale from 0 (worst) to 100 (best).
Time Frame: Day 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 100 [80 to 100]

19. Primary Outcome: Subjective Comfort With Contact Lens Wear After 6 Hours of Digital Device Use
Description: Participants rate their comfort after 6 hours of digital device use on a scale from 0 (worst) to 100 (best).
Time Frame: Day 7
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 90 [60 to 100]

20. Primary Outcome: Subjective Dryness With Contact Lens Wear After 6 Hours of Digital Device Use
Description: Participants rate their dryness after 6 hours of digital device use on a scale from 0 (worst) to 100 (best).
Time Frame: Day 7
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 90 [60 to 100]

21. Primary Outcome: Subjective Rating of Vision Clarity With Contact Lens Wear After 6 Hours of Digital Device Use
Description: Participants rate their vision clarity after 6 hours of digital device use on a scale from 0 (worst) to 100 (best).
Time Frame: Day 7
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 95 [65 to 100]

22. Primary Outcome: Subjective Comfort With Contact Lens Wear After 6 Hours of Digital Device Use
Description: Participants rate their comfort after 6 hours of digital device use on a scale from 0 (worst) to 100 (best).
Time Frame: Day 10
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 90 [75 to 100]

23. Primary Outcome: Subjective Dryness With Contact Lens Wear After 6 Hours of Digital Device Use
Description: Participants rate their dryness after 6 hours of digital device use on a scale from 0 (worst) to 100 (best).
Time Frame: Day 10
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 90 [67 to 100]

24. Primary Outcome: Subjective Rating of Vision Clarity With Contact Lens Wear After 6 Hours of Digital Device Use
Description: Participants rate their vision clarity after 6 hours of digital device use on a scale from 0 (worst) to 100 (best).
Time Frame: Day 10
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 95 [65 to 100]

25. Primary Outcome: Subjective Comfort With Contact Lens Wear After 6 Hours of Digital Device Use
Description: Participants rate their comfort after 6 hours of digital device use on a scale from 0 (worst) to 100 (best).
Time Frame: Followup visit (occurring at a single visit any day from Day 12-16)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 90 [60 to 100]

26. Primary Outcome: Subjective Dryness With Contact Lens Wear After 6 Hours of Digital Device Use
Description: Participants rate their dryness after 6 hours of digital device use on a scale from 0 (worst) to 100 (best).
Time Frame: Followup visit (occurring at a single visit any day from Day 12-16)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 90 [55 to 100]

27. Primary Outcome: Subjective Rating of Vision Clarity With Contact Lens Wear After 6 Hours of Digital Device Use
Description: Participants rate their vision clarity after 6 hours of digital device use on a scale from 0 (worst) to 100 (best).
Time Frame: Followup visit (occurring at a single visit any day from Day 12-16)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 90 [70 to 100]

28. Primary Outcome: Subjective Comfort at End of Day With Contact Lens Wear
Description: Participants rate their end of day comfort on a scale from 0 (worst) to 100 (best).
Time Frame: Day 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 100 [70 to 100]

29. Primary Outcome: Subjective Dryness at End of Day With Contact Lens Wear
Description: Participants rate their end of day dryness on a scale from 0 (worst) to 100 (best).
Time Frame: Day 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 100 [80 to 100]

30. Primary Outcome: Subjective Rating of Vision Clarity at End of Day With Contact Lens Wear
Description: Participants rate their end of day vision clarity on a scale from 0 (worst) to 100 (best).
Time Frame: Day 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 100 [80 to 100]

31. Primary Outcome: Subjective Comfort at End of Day With Contact Lens Wear
Description: Participants rate their end of day comfort on a scale from 0 (worst) to 100 (best).
Time Frame: Day 7
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 90 [60 to 100]

32. Primary Outcome: Subjective Dryness at End of Day With Contact Lens Wear
Description: Participants rate their end of day dryness on a scale from 0 (worst) to 100 (best).
Time Frame: Day 7
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 90 [60 to 100]

33. Primary Outcome: Subjective Rating of Vision Clarity at End of Day With Contact Lens Wear
Description: Participants rate their end of day rating of vision clarity on a scale from 0 (worst) to 100 (best).
Time Frame: Day 7
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 95 [65 to 100]

34. Primary Outcome: Subjective Comfort at End of Day With Contact Lens Wear
Description: Participants rate their end of day comfort on a scale from 0 (worst) to 100 (best).
Time Frame: Day 10
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 89 [60 to 100]

35. Primary Outcome: Subjective Dryness at End of Day With Contact Lens Wear
Description: Participants rate their end of day dryness on a scale from 0 (worst) to 100 (best).
Time Frame: Day 10
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 85 [40 to 100]

36. Primary Outcome: Subjective Rating of Vision Clarity at End of Day With Contact Lens Wear
Description: Participants rate their end of day vision clarity on a scale from 0 (worst) to 100 (best).
Time Frame: Day 10
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 90 [62 to 100]

37. Primary Outcome: Subjective Comfort at End of Day With Contact Lens Wear
Description: Participants rate their end of day comfort on a scale from 0 (worst) to 100 (best).
Time Frame: Followup visit (occurring at a single visit any day from Day 12-16)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 90 [60 to 100]

38. Primary Outcome: Subjective Dryness at End of Day With Contact Lens Wear
Description: Participants rate their end of day dryness on a scale from 0 (worst) to 100 (best).
Time Frame: Followup visit (occurring at a single visit any day from Day 12-16)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 88 [45 to 100]

39. Primary Outcome: Subjective Rating of Vision Clarity at End of Day With Contact Lens Wear
Description: Participants rate their end of day rating of vision clarity on a scale from 0 (worst) to 100 (best).
Time Frame: Followup visit (occurring at a single visit any day from Day 12-16)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Refit
Number analyzed (Participants) | 32
score on a scale | 90 [70 to 100]

ADVERSE EVENTS:
Time Frame: 12-16 days
Description: Regular investigator assessment. Adverse events were defined as any unfavourable and unintended sign, symptom, or disease temporarily associated with a study procedure, whether there was a causal relationship or not.
Arm/Group | Refit
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 1/32
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Refit (N=32)
Small fibre embdeed in superficial epithelium of left cornea (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was affected by the COVID-19 pandemic, which resulted in a mandated site closure to limit the spread of COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT04201639/Prot_SAP_000.pdf